CLINICAL TRIAL: NCT05089695
Title: Helmet Noninvasive Ventilation vs. Continuous Positive Airway Pressure vs. High-flow Nasal Oxygen as First-line Treatment of Acute Hypoxemic Respiratory Failure (HENIVOT2). An Open-label, Multicentre Randomized Trial
Brief Title: Helmet NIV vs. CPAP vs. High-flow Nasal Oxygen in Hypoxemic Respiratory Failure
Acronym: HENIVOT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HENIVOT2
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Failure; Hypoxemic Respiratory Failure
Keywords: Noninvasive ventilation; High-flow nasal oxygen; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Helmet Noninvasive ventilation (NIV) (Experimental): Patients in helmet noninvasive ventilation group will receive continuous helmet pressure support ventilation for at least 16 hours/day in the first 2 calendar days. Dedicated helmets for noninvasive ventilation will be applied and size will be chosen according to patient's neck circumference.
  Each patient will be connected to a mechanical ventilator ventilator through a bitube circuit with no humidification.
  The ventilator will be set in PSV-NIV mode, with the following suggested settings [34-38]:
  1. initial pressure support=12 cmH2O and adequate to permit a peak inspiratory flow of 100 l/min;
  2. positive end-expiratory pressure=12 cmH2O.
  3. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  4. Inspiratory flow trigger = 2 l/min or according to the practice of each institution;
  5. fastest pressurization time;
  6. expiratory trigger: 10-50% of the maximum inspiratory flow, eventually modified to avoid double triggering;
  7. maximum inspiratory time 1.2 second.
  Interventions: Device: Noninvasive respiratory support
- Helmet continuous airway pressure (CPAP) (Experimental): Patients in CPAP group will receive continuous helmet CPAP for at least 16 hours/day in the first 2 calendar days. Continuous CPAP without interruptions will be strongly encouraged in the first 48 hours of treatment. Dedicated helmets for noninvasive ventilation will be applied and size will be chosen according to patient's neck circumference.
  Treatment will be delivered through a high-flow generator. The following settings will be applied:
  1. Continuous air flow>45 l/min.
  2. Bi-tube circuit with no humidification, Y-piece with heat and moisture exchanger, or active heating and humidification with humidification chamber temperature set at 31 °C, 34 °C or 37 °C according to patients' comfort.
  3. Expiratory positive end-expiratory pressure valve set to achieve PEEP=12 cmH2O.
  4. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  Interventions: Device: Noninvasive respiratory support
- High-flow nasal oxygen (Active Comparator): Initial set flow will be 50-60 l/min and flows will be decreased. in case of intolerance and/or according to patients' requirements: flows≥30 L/min will be mandatory in all enrolled patients. Humidification chamber will be set at 31 °C, 34 °C or 37 °C according to patient's comfort. FiO2 will be titrated to obtain an SpO2≥92% and ≤98%.
  Weaning the patient from high-flow will be considered only after 48 hours from enrolment and will be discouraged until the patients is considered for ICU discharge.
  Interventions: Device: Noninvasive respiratory support

INTERVENTIONS:
Device: Noninvasive respiratory support — Treatment of acute hypoxemic respiratory failure

SUMMARY:
Multicenter, open label, three-arm randomized trial to assess the effect of helmet noninvasive ventilation vs. helmet continuous positive airway pressure vs. high-flow nasal oxygen on the rate of endotracheal intubation of patients with acute moderate-to-severe hypoxemic respiratory failure

DETAILED DESCRIPTION:
The optimal initial management of acute hypoxemic respiratory failure is uncertain. Helmet noninvasive ventilation and high-flow nasal oxygen appear as the most promising techniques in this setting. Recently, the first head-to-head randomized trial compared first-line continuous treatment with helmet pressure support ventilation with specific settings (PEEP=12 cmH2O pressure and pressure support=10-12 cmH2O) vs. high-flow nasal oxygen alone in patients with moderate-to-severe hypoxemic respiratory failure. Results showed no significant inter-group difference in the days free of respiratory support at 28 days, but lower intubation rate and increased 28-day invasive ventilation-free days in the helmet group. Use of helmet noninvasive ventilation is less frequent than use of helmet continuous positive airway pressure, which is simpler to use.

The investigators designed an open-label, multicentre randomized trial to assess the effect of helmet pressure support ventilation and continuous airway pressure as compared to high-flow nasal oxygen on the intubation rate of patients with moderate-to-severe hypoxemic respiratory failure in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Acute symptoms of respiratory failure PaO2/FiO2 ratio ≤ 200; PaCO2≤45mmHg; Absence of history of chronic respiratory failure or moderate to severe cardiac insufficiency (NYHA>2 or left ventricular ejection fraction<50%); Informed consent

Patients that have already received NIV, CPAP continuously for more than 24 hours before the screening visit will be excluded.

Other Exclusion Criteria:

* Pregnancy;
* Exacerbation of asthma or chronic obstructive pulmonary disease;
* Hypercapnia (PaCO2>45 mmHg) with or without respiratory acidosis;
* More than 2 organ failures, including the lung.
* Documented pneumothorax;
* Clinical diagnosis of Cardiogenic pulmonary edema;
* Haemodynamic instability (Systolic blood pressure<90 mmHg or mean arterial pressure<65mmHg) and/or lactic acidosis (lactate>5 mmol/L) and/or clinically diagnosed Shock requiring administration of vasoactive agents (norepinephrine>0.1 mcg/Kg/min);
* Metabolic Acidosis (pH <7.30 with normal- or hypo-carbia);
* Chronic kidney failure requiring dialysis before ICU admission;
* Chronic hypoxemic respiratory failure requiring long-term oxygen therapy;
* Altered neurological status that requires immediate intubation and/or making the patient uncooperative;
* Urgent need for endotracheal intubation, according to the decision of the attending physician;
* Do not intubate order;
* Decision of withdrawal of life-sustaining therapy;
* Thoracic or abdominal surgery in the previous 7 days;
* Any condition that makes the patient very likely to require endotracheal intubation due to a reason different from respiratory failure;
* Recent head surgery or anatomy that prevent the application of helmet or HFNC to patient's face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Endotracheal intubation | 28 days
  The proportion of patients requiring endotracheal intubation according to predefined criteria

SECONDARY OUTCOMES:
Days free of invasive mechanical ventilation at day 28 | 28 days
  The number of days in which patients do not receive mechanical ventilation within 28 days from randomization
Days free of invasive mechanical ventilation at day 60 | 60 days
  The number of days in which patients do not receive mechanical ventilation within 60 days from randomization
Days free of invasive mechanical ventilation at day 90 | 90 days
  The number of days in which patients do not receive mechanical ventilation within 60 days from randomization
Rate of In-intensive care unit mortality | 90 days
  All-cause mortality, assessed at the discharge from the intensive care unit
Rate of In-hospital care unit mortality | 90 days
  All-cause mortality, assessed at the discharge from the hospital
Rate of 90-day mortality | 90 days
  All-cause 90-day mortality
90-day ICU free days | 90 days
  The days not spent in the intensive care unit by the patient on a 90-day basis
90-day hospital free days | 90 days
  The days not spent in the hospital by the patient on a 90-day basis
Incidence of pneumonia | 90 days
  Incidence of pneumonia, diagnosed after the treatment start and during the ICU stay
Incidence of shock | 90 days
  Incidence of shock, diagnosed after treatment start and during the ICU stay
Incidence of barotrauma | 90 days
  Incidence of barotrauma, defined as pneumothorax o pneumomediastinum after treatment start and during the ICU stay

OTHER OUTCOMES:
Safety endpoint-causes of endotracheal intubation | 28 days
  Among patients meeting the primary endpoint, the cause of noninvasive treatment failure (as defined by the predefined intubation criteria)
Safety endpoint-time to treatment failure | 28 days
  In patients meeting the primary endpoint, the time (hours) from randomization to intubation

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Luca Grieco, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS; Massimo Antonelli, MD, Study Chair — Fondazione Policlinico A. Gemelli IRCCS
Locations (1):
- Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be made available by the principal investigator upon a reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: With publication the results
Access Criteria: Individual data will be made available by the principal investigator upon a reasonable request